CLINICAL TRIAL: NCT02303899
Title: A Phase II Study of the Combination of Gemcitabine and Imatinib Mesylate in Pemetrexed-pretreated Patients With Malignant Pleural Mesothelioma
Brief Title: Combination of Gemcitabine and Imatinib Mesylate in Pemetrexed-pretreated Patients With Pleural Mesothelioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2014-002
Record Dates: First submitted 2014-11-19; First posted 2014-12-01 (Estimated); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Mesothelioma, Malignant
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Gemcitabine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine & Imatinib mesylate (Experimental): Gemcitabine 1000 mg/m2, i.v., days 3 and 10 of a 21-days schedule; Imatinib mesylate 400 mg/die orally on days 1-5 and 8-12 of a 21-days schedule.
  Interventions: Drug: Gemcitabine; Drug: Imatinib mesylate

INTERVENTIONS:
Drug: Gemcitabine — infusion drug
  Other Names: Gemzar
Drug: Imatinib mesylate — oral drug
  Other Names: Glivec

SUMMARY:
This is a phase II, monocentric study of the combination of gemcitabine and imatinib mesylate in pemetrexed-pretreated patients with MPM expressing PDGFR-beta and/or C-kit by Immunohistochemistry (IHC). Treatment will be done until disease progression, or patient refusal or withdrawal of patient consent, or unacceptable toxicity

DETAILED DESCRIPTION:
Pemetrexed-pretreated patients with MPM expressing PDGFR-beta and/or C-kit by IHC will receive chemotherapy as follow :

* Gemcitabine 1000 mg/m2, i.v., days 3 and 10 of a 21-days schedule;
* Imatinib mesylate 400 mg/die orally on days 1-5 and 8-12 of a 21-days schedule.

Treatment repeats every 21 days in the absence of disease progression, patient refusal or withdrawal of patient consent, or unacceptable toxicity.

The molecular profile of patients enrolled will be evaluated with Ion Personal Genome Machine (PGM) Torrent Next-generation Sequencing platform in order to individuate potential predictive biomarkers and to improve the understanding of the molecular biology of these rare tumors. A correlation among the molecular profiles identified, clinical characteristics, and survival data of patients will be done

ELIGIBILITY:
Inclusion Criteria:

1. Age of > 18 years.
2. Histologically proven malignant mesothelioma of the pleura or of the peritoneum, expressing PDGFR-beta and/or C-kit by immunohistochemistry.
3. Locally advanced disease, unsuitable for curative surgical resection, or metastatic disease.
4. Confirmed progression of the disease according to modified RECIST-criteria, documented after a pemetrexed-based chemotherapy.
5. Eastern Cooperative Oncology group (ECOG) Performance Status of 0, 1 or 2.
6. Life expectancy of at least 3 months.
7. Written informed consent.

Exclusion Criteria:

1. Co-existing tumors of different histologic origin, except non melanomatous localized skin cancer and/or in situ cervical carcinoma.
2. A history of earlier tumors of different histologic origin being in complete remission for less than 5 years.
3. Unresolved toxicity from prior antitumor treatment(s).
4. Primary peritoneal mesothelioma.
5. Any of the following abnormal baseline hematological values:

   * Hb < 9 g/dL
   * White blood count (WBC) < 3 x 109/L
   * Neutrophils < 1.5 x 109/L
   * Platelets < 100 x 109/L
   * Serum bilirubin > 2.5 mg/dL
   * Alanine transaminase (ALAT) and Aspartate transaminase (ASAT) > 3 x upper normal limit (UNL) (unless due to liver metastases)
   * Serum creatinine > 1.5 mg/dL.
6. Symptomatic and/or unstable pre-existing brain metastases. To be enrolled in the study, subjects must have confirmation of stable disease by MRI or computer tomography (CT) scan within 4 weeks from day 1 of cycle 1 of treatment and have central nervous system (CNS) metastases well controlled by steroids, anti - epileptics or other symptom-relieving medications.
7. Clinically relevant cardiovascular disease, i.e., myocardial infarction or other severe coronary artery diseases within the prior 6 months, cardiac arrythmia requiring medication, uncontrolled hypertension, overt cardiac failure or non compensated chronic heart disease in New York Heart Association (NYHA) class II or more.
8. History of psychiatric disabilities, potentially interfering with the capability of giving adequate informed consent.
9. Pregnant or lactating women or inability/unwillingness to practice a medically approved method of contraception during study period (including 3 months following the end of treatment)
10. Uncontrolled active infections.
11. Any condition which, in the judgement of the Investigator, would place the patient at undue risk or interfere with the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
anti-tumor activity of Imatinib mesylate in combination with Gemcitabine | 12 weeks
  assess the anti-tumor activity of Imatinib mesylate in combination with Gemcitabine, in terms of 3-months progression-free survival (PFS) rate

SECONDARY OUTCOMES:
anti-tumor activity of Imatinib mesylate in combination with Gemcitabine in terms of Response Evaluation Criteria In Solid Tumors (RECIST) criteria | 16 weeks
  assess anti-tumor activity of Imatinib Mesylate (IM) in combination with GEM, in terms of objective response rate according to RECIST criteria (Modified RECIST criteria for MPM), and duration of response
anti-tumor activity of Imatinib mesylate in combination with Gemcitabine in terms of overall survival (OS). | 30 months
  assess anti-tumor activity of IM in combination with GEM, in terms of overall survival (OS).
safety profile of the combination according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3 | 16 weeks
  determine the safety profile of the combination according to the National Cancer Institute Common Toxicity Criteria (NCI-CTC) version 3
molecular profile of patients | baseline
  evaluate the molecular profile of patients enrolled with Ion PGM Torrent Next-generation Sequencing platform correlating the molecular profiles identified with clinical characteristics and survival data of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No
not planned

REFERENCES:
- [Background] Vogelzang NJ, Rusthoven JJ, Symanowski J, Denham C, Kaukel E, Ruffie P, Gatzemeier U, Boyer M, Emri S, Manegold C, Niyikiza C, Paoletti P. Phase III study of pemetrexed in combination with cisplatin versus cisplatin alone in patients with malignant pleural mesothelioma. J Clin Oncol. 2003 Jul 15;21(14):2636-44. doi: 10.1200/JCO.2003.11.136. PMID 12860938
- [Background] Ceresoli GL, Zucali PA, Favaretto AG, Grossi F, Bidoli P, Del Conte G, Ceribelli A, Bearz A, Morenghi E, Cavina R, Marangolo M, Parra HJ, Santoro A. Phase II study of pemetrexed plus carboplatin in malignant pleural mesothelioma. J Clin Oncol. 2006 Mar 20;24(9):1443-8. doi: 10.1200/JCO.2005.04.3190. PMID 16549838
- [Background] Castagneto B, Botta M, Aitini E, Spigno F, Degiovanni D, Alabiso O, Serra M, Muzio A, Carbone R, Buosi R, Galbusera V, Piccolini E, Giaretto L, Rebella L, Mencoboni M. Phase II study of pemetrexed in combination with carboplatin in patients with malignant pleural mesothelioma (MPM). Ann Oncol. 2008 Feb;19(2):370-3. doi: 10.1093/annonc/mdm501. Epub 2007 Dec 20. PMID 18156144
- [Background] Santoro A, O'Brien ME, Stahel RA, Nackaerts K, Baas P, Karthaus M, Eberhardt W, Paz-Ares L, Sundstrom S, Liu Y, Ripoche V, Blatter J, Visseren-Grul CM, Manegold C. Pemetrexed plus cisplatin or pemetrexed plus carboplatin for chemonaive patients with malignant pleural mesothelioma: results of the International Expanded Access Program. J Thorac Oncol. 2008 Jul;3(7):756-63. doi: 10.1097/JTO.0b013e31817c73d6. PMID 18594322
- [Background] Ceresoli GL, Zucali PA, Gianoncelli L, Lorenzi E, Santoro A. Second-line treatment for malignant pleural mesothelioma. Cancer Treat Rev. 2010 Feb;36(1):24-32. doi: 10.1016/j.ctrv.2009.09.003. Epub 2009 Oct 29. PMID 19879055
- [Background] Pietras K, Ostman A, Sjoquist M, Buchdunger E, Reed RK, Heldin CH, Rubin K. Inhibition of platelet-derived growth factor receptors reduces interstitial hypertension and increases transcapillary transport in tumors. Cancer Res. 2001 Apr 1;61(7):2929-34. PMID 11306470
- [Background] Pietras K, Rubin K, Sjoblom T, Buchdunger E, Sjoquist M, Heldin CH, Ostman A. Inhibition of PDGF receptor signaling in tumor stroma enhances antitumor effect of chemotherapy. Cancer Res. 2002 Oct 1;62(19):5476-84. PMID 12359756
- [Background] Pietras K, Stumm M, Hubert M, Buchdunger E, Rubin K, Heldin CH, McSheehy P, Wartmann M, Ostman A. STI571 enhances the therapeutic index of epothilone B by a tumor-selective increase of drug uptake. Clin Cancer Res. 2003 Sep 1;9(10 Pt 1):3779-87. PMID 14506171
- [Background] Garlepp MJ, Leong CC. Biological and immunological aspects of malignant mesothelioma. Eur Respir J. 1995 Apr;8(4):643-50. PMID 7664867
- [Background] Langerak AW, van der Linden-van Beurden CA, Versnel MA. Regulation of differential expression of platelet-derived growth factor alpha- and beta-receptor mRNA in normal and malignant human mesothelial cell lines. Biochim Biophys Acta. 1996 Feb 7;1305(1-2):63-70. doi: 10.1016/0167-4781(95)00196-4. PMID 8605252
- [Background] Pogrebniak HW, Lubensky IA, Pass HI. Differential expression of platelet derived growth factor-beta in malignant mesothelioma: a clue to future therapies? Surg Oncol. 1993 Aug;2(4):235-40. doi: 10.1016/0960-7404(93)90012-n. PMID 8252214
- [Background] Klominek J, Baskin B, Hauzenberger D. Platelet-derived growth factor (PDGF) BB acts as a chemoattractant for human malignant mesothelioma cells via PDGF receptor beta-integrin alpha3beta1 interaction. Clin Exp Metastasis. 1998 Aug;16(6):529-39. doi: 10.1023/a:1006542301794. PMID 9872600
- [Background] Sawyers C. Targeted cancer therapy. Nature. 2004 Nov 18;432(7015):294-7. doi: 10.1038/nature03095. PMID 15549090
- [Background] Shih AH, Holland EC. Platelet-derived growth factor (PDGF) and glial tumorigenesis. Cancer Lett. 2006 Feb 8;232(2):139-47. doi: 10.1016/j.canlet.2005.02.002. Epub 2005 Aug 31. PMID 16139423
- [Background] Yu J, Ustach C, Kim HR. Platelet-derived growth factor signaling and human cancer. J Biochem Mol Biol. 2003 Jan 31;36(1):49-59. doi: 10.5483/bmbrep.2003.36.1.049. PMID 12542975
- [Background] Johnson MD, Okedli E, Woodard A, Toms SA, Allen GS. Evidence for phosphatidylinositol 3-kinase-Akt-p7S6K pathway activation and transduction of mitogenic signals by platelet-derived growth factor in meningioma cells. J Neurosurg. 2002 Sep;97(3):668-75. doi: 10.3171/jns.2002.97.3.0668. PMID 12296652
- [Background] Porta C, Mutti L, Tassi G. Negative results of an Italian Group for Mesothelioma (G.I.Me.) pilot study of single-agent imatinib mesylate in malignant pleural mesothelioma. Cancer Chemother Pharmacol. 2007 Jan;59(1):149-50. doi: 10.1007/s00280-006-0243-4. Epub 2006 Apr 25. No abstract available. PMID 16636799
- [Background] Roberts F, Harper CM, Downie I, Burnett RA. Immunohistochemical analysis still has a limited role in the diagnosis of malignant mesothelioma. A study of thirteen antibodies. Am J Clin Pathol. 2001 Aug;116(2):253-62. doi: 10.1309/XL6K-8E62-9FLD-V8Q8. PMID 11488073
- [Background] George D. Platelet-derived growth factor receptors: a therapeutic target in solid tumors. Semin Oncol. 2001 Oct;28(5 Suppl 17):27-33. PMID 11740804
- [Background] Taylor JR, Brownlow N, Domin J, Dibb NJ. FMS receptor for M-CSF (CSF-1) is sensitive to the kinase inhibitor imatinib and mutation of Asp-802 to Val confers resistance. Oncogene. 2006 Jan 5;25(1):147-51. doi: 10.1038/sj.onc.1209007. PMID 16170366
- [Background] Mathy A, Baas P, Dalesio O, van Zandwijk N. Limited efficacy of imatinib mesylate in malignant mesothelioma: a phase II trial. Lung Cancer. 2005 Oct;50(1):83-6. doi: 10.1016/j.lungcan.2005.04.010. PMID 15951053
- [Background] Bertino P, Porta C, Barbone D, Germano S, Busacca S, Pinato S, Tassi G, Favoni R, Gaudino G, Mutti L. Preliminary data suggestive of a novel translational approach to mesothelioma treatment: imatinib mesylate with gemcitabine or pemetrexed. Thorax. 2007 Aug;62(8):690-5. doi: 10.1136/thx.2006.069872. Epub 2007 Feb 20. PMID 17311837
- [Background] Bertino P, Piccardi F, Porta C, Favoni R, Cilli M, Mutti L, Gaudino G. Imatinib mesylate enhances therapeutic effects of gemcitabine in human malignant mesothelioma xenografts. Clin Cancer Res. 2008 Jan 15;14(2):541-8. doi: 10.1158/1078-0432.CCR-07-1388. PMID 18223230
- [Background] George S, Desai J, Paul Eder J, Manola J, Ryan DP, Appleman LJ, Demetri GD. Selective kinase inhibition with daily imatinib intensifies toxicity of chemotherapy in patients with solid tumours. Eur J Cancer. 2006 May;42(7):864-70. doi: 10.1016/j.ejca.2005.12.010. Epub 2006 Feb 28. PMID 16503137
- [Background] Ali Y, Lin Y, Gharibo MM, Gounder MK, Stein MN, Lagattuta TF, Egorin MJ, Rubin EH, Poplin EA. Phase I and pharmacokinetic study of imatinib mesylate (Gleevec) and gemcitabine in patients with refractory solid tumors. Clin Cancer Res. 2007 Oct 1;13(19):5876-82. doi: 10.1158/1078-0432.CCR-07-0883. PMID 17908982
- [Background] Byrne MJ, Nowak AK. Modified RECIST criteria for assessment of response in malignant pleural mesothelioma. Ann Oncol. 2004 Feb;15(2):257-60. doi: 10.1093/annonc/mdh059. PMID 14760119
- See also: 27) National Cancer Institute. Common toxicity criteria manual, version 3.0, July 16, 2003. — http://ctep.cancer.gov/reporting/ctc.html